CLINICAL TRIAL: NCT01217736
Title: Direct Renin Inhibition and the Kidney
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vitae Pharmaceuticals, Inc. (Industry)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VTP-27999-005; 2010P001281 (Other: Partners Healthcare System)
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Renal Function
MeSH Terms: interventions — aliskiren; methyl (2-((3-chlorophenyl)(1-((2-(methylamino)-3-(tetrahydro-2H-pyran-3-yl)propyl)carbamoyl)piperidin-3-yl)methoxy)ethyl)carbamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VTP-27999 (Experimental)
  Interventions: Drug: VTP-27999
- aliskiren (Active Comparator)
  Interventions: Drug: aliskiren
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aliskiren — single dose, tablet
  Other Names: Tekturna
  Arms: aliskiren
Drug: placebo — single dose, tablet
  Arms: placebo
Drug: VTP-27999 — single dose, tablet
  Arms: VTP-27999

SUMMARY:
The objective of the study is to determine the magnitude of the effect of direct renin inhibition by VTP-27999 on renal plasma flow and kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female, 18-75 years of age
* Female subjects must be postmenopausal or surgically sterilized. Postmenopausal females must have had no regular menstrual bleeding for at least one (1) year prior to initial dosing. Menopause will be confirmed by plasma serum FSH level at screening between 23.0-116.3 mIU/ml. Female subjects who report surgical sterilization must have had the procedure at least six (6) months prior to initial dosing.
* Male subjects, able to father a child, must be willing to use approved birth control methods for 2 weeks following completion of study.

Exclusion Criteria:

* Subjects under 18 and subjects over 75 years
* Diabetes Mellitus and/or kidney disease
* Myocardial infarction, stroke, or cardiovascular revascularization/angioplasty within the last 6 months
* Unstable angina pectoris or CAD requiring treatment with an excluded concomitant medication
* History of/or symptoms consistent with congestive heart failure
* Hypertension
* History of left ventricular ejection fraction < 45%
* Current smokers or nicotine patch
* Pregnant or lactating females
* Cancer or any life threatening illness with expected death within 2 years or by completion of the study
* Serum creatinine >1.4 mg/dl
* Serum potassium <3.5 or >5.2 mmol/L without medication
* Serum albumin < 2.0 g/dL
* Hemoglobin < 11.5 g/dL or Hematocrit < 34%
* Any serum AST >/= 60 or ALT >/= 75 IU/L
* Use of any prescription drugs which may affect the renin-angiotensin-aldosterone system or with known effect on renal hemodynamics are not allowed within 10 days prior to dosing or during the study
* Use of CYP3A4 inhibitors (e.g. Diltiazem, Ketoconazole, Nifedipine, or Verapamil)
* Use of any prescription medication is prohibited within 14 days (or, if known, for at least 5 half-lives, if longer) prior to dosing, unless approved by both the Investigator and the Sponsor
* Use of any over-the-counter (OTC) medication, including herbal products, is prohibited within the 14 days prior to dosing, unless approved by both the Investigator and the Sponsor
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing
* A known hypersensitivity or contraindication to the study drugs (Aliskiren) or drugs similar to the study drugs or PAH, and inulin
* Any surgical or medical condition which alters absorption, distribution, metabolism or excretion of drugs or which may jeopardize the patient subject during this study, including gastric bypass
* History of drug or alcohol abuse within the 12 months prior to dosing, or evidence of such abuse as indicated by past medical history
* Acute infections and/or significant illness within 3 weeks of planned enrollment into this study
* Any medical condition in the investigator's opinion, which renders the subject unable to complete the study or which would produce significant risk to the subject
* Administration of any other investigational drug within 30 days of planned dosing in the study
* Poor intravenous (IV) access as determined by the study staff

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
renal plasma flow | pre-dose to 6 hours post-dose
  as measured by PAH clearance

SECONDARY OUTCOMES:
glomerular filtration rate | pre-dose to 6 hours post-dose
RAAS pathway biomarkers | pre-dose to 24 hours post-dose
  renin, prorenin, plasma renin activity, ang II
VTP-27999 concentrations | pre-dose to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Norman K Hollenberg, MD, PhD, Principal Investigator — Brigham and Women's Hospital, Boston, MA
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Barkoudah E, Danser AHJ, van Thiel BS, Fisher NDL, Gregg R, Hollenberg NK. Journal of the American Society of Hypertension 9(4)
- [Result] Barkoudah E, van Thiel BS, Fisher ND, Gregg RA, Danser AH, Moukarbel GV, Hollenberg NK. Maximum renal responses to renin inhibition in healthy study participants: VTP-27999 versus aliskiren. J Hypertens. 2016 May;34(5):935-41. doi: 10.1097/HJH.0000000000000860. PMID 26882043
- See also: maximum renal responses in healthy study participants: VTP-27999 versus aliskiren — http://www.ncbi.nlm.nih.gov/pubmed/26882043